CLINICAL TRIAL: NCT07028476
Title: NPS-LDA - New Care Pathway Using Automated Dynamic Laximetry
Brief Title: New Care Pathway Using Automated Dynamic Laximetry
Acronym: NPS-LDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC23_0427
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Knee Sprain; Automated Dynamic Laximetry (ADL); Care Pathway; MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pds-IRM (Experimental)
  Interventions: Procedure: MRI
- Pds-LDA (Active Comparator)
  Interventions: Procedure: Automated Dynamic Laximetry

INTERVENTIONS:
Procedure: Automated Dynamic Laximetry — Patients are prescribed a Zimmer splint to immobilize the injured limb, and referred to a referring sports physician at the investigating center to perform the LDA as a confirmatory examination (complementary test). Patients arrange their appointment with the sports physician as soon as possible.
  Arms: Pds-LDA
Procedure: MRI — In the control arm, and in line with standard practice, patients with a suspected ACL injury are prescribed a Zimmer splint to immobilize the injured limb, an MRI as a confirmatory examination, and a consultation with the doctor of their choice. Following the MRI, patients arrange their appointments according to the usual care pathway for their pathology.
  Arms: Pds-IRM

SUMMARY:
Today, in the event of a knee sprain with suspected cruciate ligament damage, magnetic resonance imaging (MRI) is generally prescribed to confirm or refute the diagnosis and assess its severity. Once the MRI has been performed, the patient's care is organized by the doctor of his or her choice, depending on the diagnosis.

Previous studies have shown that Automated Dynamic Laximetry (ADL) performs identically to MRI in helping to diagnose a knee sprain as a complementary examination and in assessing its severity. Performing LDA at the start of the patient's care pathway, i.e. immediately after the emergency room visit for a suspected severe sprain, could bring significant benefits by shortening the diagnostic confirmation time and consequently the immobilization period, and by reducing the cost of care compared with the conventional MRI-based care pathway. The new LDA-based care pathway would enable MRI to be reserved for very specific cases, such as the scheduling of surgery for suspected meniscus or osteochondral lesions, as currently recommended by the HAS.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to an emergency department participating in the study
* Age ≥ 18 years
* Consulted following knee trauma and whose clinical examination leads to the suspicion of a partial or complete ACL lesion without bone fracture (supporting radiograph).
* Signed consent to participate in the study
* Affiliated to a social security scheme

Exclusion Criteria:

* Contraindication to MRI (pacemaker fitted before 2010) or LDA;
* Indication for emergency or semi-emergency trauma surgery (within 3 weeks: suspected unstable meniscal lesion, fracture, etc.).
* Impossible follow-up or patient's refusal of follow-up in the investigating center's sports medicine department;
* Poor understanding of the French language
* Pregnant (known or suspected pregnancy), breast-feeding or parturient woman;
* Person deprived of liberty by judicial or administrative decision;
* Person under compulsory psychiatric care;
* Person subject to a legal protection measure
* Person unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
KOOS questionnaire | Inclusion, 1 month, 3 months, 6 months and 12 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is used to assess immediate and long-term patient outcomes following knee injury. Five outcomes are assessed by the self-administered KOOS: pain, symptoms, activities of daily living, sports and recreational function, and knee-related quality of life. KOOS meets basic standards for outcome measures and can be used to assess the evolution of the knee injury and the effectiveness of treatment. KOOS is patient-administered, has an easy-to-use format and takes around 10 minutes to complete.
EQ-5D-5L questionnaire | Inclusion, 1 month, 3 months, 6 months and 12 months
  The EQ5D-5L question listings are designed to analyze quality of life across 5 themes (mobility, personal autonomy, daily activities, pain/discomfort, anxiety/depression and health assessment).
Tegner activity scale | Inclusion, 1 month, 3 months, 6 months and 12 months
  The Tegner Activity Scale is a numerical scale ranging from 0 to 10, with each value indicating the ability to perform specific activities. Higher scores represent participation in higher-level activities.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Angers, Angers
  - CH LAVAL, Laval
  - Chu Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No